CLINICAL TRIAL: NCT02725931
Title: Impact of Feedback on Physical Activity Levels and Health-related Outcomes of Patients With COPD During Pulmonary Rehabilitation
Brief Title: Impact of Feedback on Physical Activity and Health-related Outcomes During Pulmonary Rehabilitation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SFRH /BD/81328/2011
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease; COPD; Pulmonary rehabilitation; Physical activity; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activity group (Experimental): Pulmonary rehabilitation plus physical activity intervention
  Interventions: Behavioral: Pulmonary rehabilitation (PR) plus PA-focused intervention

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation (PR) plus PA-focused intervention — Patients will enrol in a 12-week PR program comprising exercise training (3 times per week) and psychosocial support and education sessions (once a week). Patients will also have their PA levels monitored on weeks (W) 1, 7 and 12 and receive feedback in the following weeks.

SUMMARY:
The aim of this study is to investigate whether providing feedback on physical activity (PA) levels to patients with Chronic Obstructive Pulmonary Disease (COPD) is feasible and enhances daily PA and health-related outcomes during pulmonary rehabilitation (PR).

Patients will participate in a 12-week PR program and a PA-focused intervention. Patients' daily PA will be monitored during the first (W1), seventh (W7) and 12th (W12) weeks of the PR program using the activity monitors GT3X+ (ActiGraph, Pensacola, FL) and feedback will be given to them in the following weeks. Each participant will also receive individualised recommendations to improve or maintain their PA levels, based on the results of the previous week.

It is expected that, by receiving individualised feedback and goals regarding their PA levels during the PR program, patients with COPD will become more active and improve their health-related outcomes.

DETAILED DESCRIPTION:
Patients with Chronic Obstructive Pulmonary Disease (COPD) present lower levels of physical activity (PA), which have been associated with adverse outcomes including increased healthcare utilisation and reduced survival. Thus, improving PA levels has become one of the main goals of COPD research.

Pulmonary rehabilitation (PR) is a cornerstone of COPD management with well-documented effects on exercise capacity and quality of life. However, its effects in increasing patients' physical activity (PA) levels are limited. Previous research has suggested that PR with PA monitoring and feedback may be a suitable approach to increase and/or maintain patients' PA levels.

Patients with COPD will participate in a 12-week PR program plus a PA-focused intervention. Daily PA will be measured using activity monitors GT3X+ (ActiGraph, Pensacola, FL) on weeks (W) 1, 7 and 12 and feedback will be given to participants in the following weeks regarding: daily steps; time spent in sedentary, light and moderate-to-vigorous (MVPA) intensity activities.

The impact of the intervention will be explored using a mixed-methods approach.

Assessments will be conducted immediately before (W1) and after (W12) the PR program. Breathlessness, exercise capacity, functional balance, peripheral muscle strength and health-related quality of life will be assessed in both time points.

Descriptive statistics will be used to characterise the sample. To analyse changes in outcome measures, data from the two time points will be compared. Correlations between PA data and health-related outcomes will be performed at W1 and using the change scores (i.e., W12-W1).

Patients will also be invited to attend focus groups after the intervention to assess their perspectives about the use of activity monitors and the feedback given.

This is a pilot study which will inform the main study (including the sample size calculation).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria
* ≥ 18 years old
* clinical stability for 1 month prior to the study (no hospital admissions or exacerbations)

Exclusion Criteria:

* presence of severe psychiatric, neurologic or musculoskeletal conditions and/or unstable cardiovascular disease
* participation in regular exercise prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in physical activity levels | weeks 1, 7 and 12
  Physical activity data will be collected using a triaxial accelerometer. Number of steps per day and time spent in sedentary, light and moderate-to-vigorous intensity activities will be assessed. Time spent in different postures (i.e., standing, sitting and lying) will also be determined.

SECONDARY OUTCOMES:
Change in exercise capacity | immediately before (week 1) and after (week 12) the PR program
  Exercise tolerance will be assessed with the 6-minute walk test, following the American Thoracic Society guidelines. The maximal distance walked during 6 minutes and the associated respiratory symptoms will be collected.
Change in peripheral muscle strength | immediately before (week 1) and after (week 12) the PR program
  Isometric muscle strength of the upper and lower limbs will be assessed with the 10-RM following the American College of Sports Medicine guidelines.
Change in activities limitation resulting from breathlessness | immediately before (week 1) and after (week 12) the PR program
  The Modified British Medical Research Council questionnaire comprises five grades (statements) in a scale from 0 to 4, with higher grades indicating greater perceived respiratory limitation.
Change in functional balance | immediately before (week 1) and after (week 12) the PR program
  The Timed Up and Go (TUG) test is a functional balance test in which the time needed to perform the test is recorded.
Change in health-related quality of life | immediately before (week 1) and after (week 12) the PR program
  The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure quality of life in patients with chronic lung disease. It has 3 domains: symptoms, activities and impact. Higher scores indicate poorer quality of life.
Patients' perspectives about the intervention | Immediately after the PR program (week 12)
  Semi-structured focus group interviews will be conducted with patients to explore their perspectives about the use of activity monitors and the feedback given.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, PhD, Principal Investigator — Aveiro University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cruz J, Brooks D, Marques A. Impact of feedback on physical activity levels of individuals with chronic obstructive pulmonary disease during pulmonary rehabilitation: A feasibility study. Chron Respir Dis. 2014 Nov;11(4):191-8. doi: 10.1177/1479972314552280. Epub 2014 Oct 2. PMID 25278009